CLINICAL TRIAL: NCT06226246
Title: Evaluation of Effectiveness of Virtual Reality-based Dispatcher Assisted Cardiopulmonary Resuscitation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 0420232290
Record Dates: First submitted 2024-01-03; First posted 2024-01-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest
Keywords: CPR education; Virtual reality
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HEROS VR (Experimental): Trainee trained by HEROS VR CPR training program
  Interventions: Behavioral: HEROS VR CPR training program
- Conventional HEROS (Active Comparator): Trainee trained by conventional HEROS CPR training program
  Interventions: Behavioral: Conventional HEROS CPR training program

INTERVENTIONS:
Behavioral: HEROS VR CPR training program — HEROS VR training program which combined video training and VR session
  Arms: HEROS VR
Behavioral: Conventional HEROS CPR training program — Conventional HEROS training program using video learning
  Arms: Conventional HEROS

SUMMARY:
This study aims to compare the effect of conventional cardiopulmonary resuscitation (CPR) training and CPR training with added virtual reality (VR) on trainee self-efficacy.

DETAILED DESCRIPTION:
This study aims to compare the conventional cardiopulmonary resuscitation (CPR) training program (HEROS CPR training program) with the HEROS VR (virtual reality) CPR training program to which the newly developed VR curriculum was added. The experimental group is the HEROS VR training group, and CPR training is conducted for approximately 60 minutes for 6 to 8 trainees per training. At the start and the end of the training, students are taught about cardiac arrest, recognition of emergency situations, and reporting to 119 by watching VR, and in the middle part, they practice chest compressions by watching conventional HEROS video. The control group is the existing HEROS training group. To control variables, the number of trainees per training was limited to 6 to 8, and the existing video-based CPR training was implemented. The investigators will conduct a Modified Basic Resuscitation Skills Self-Efficacy scale survey before and after training to compare the difference in the improvement of trainees' self-efficacy evaluation of CPR after CPR training in the HEROS VR curriculum and the existing HEROS curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Non-medical personnel aged 18~65

Exclusion Criteria:

* Who have received CPR training within the past 1 year.
* For whom it is difficult to wear the VR equipment due to a history of side effects or problems such as head trauma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-23 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Modified Basic Resuscitation Skills Self-Efficacy scale | Immediately before training and immediately after the training program
  Modified Basic Resuscitation Skills Self-Efficacy scale (Modified BRS-SES):
  The scale consists of 8 questionnaires with a 5-point Likert scale. After aggregating the scores, the score is converted to a scale of 100 points, with a minimum score of 20 and a maximum of 100. A higher score indicates a higher level of self-efficacy.

SECONDARY OUTCOMES:
System Usability Scale | Immediately after the VR training program
  System Usability Scale for VR device:
  The scale consists of 10 item questionnaire with five response options from strongly agree to strongly disagree. The results of the 10 questions are aggregated and converted to a score out of 100. The higher the score the higher the usability.

CONTACTS AND LOCATIONS:
Overall Officials: STEPHEN LEE, MD, MA, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park GJ, Kong SYJ, Song KJ, Shin SD, Kim TH, Ro YS, Myklebust H, Birkenes TS. The Effectiveness of a New Dispatcher-Assisted Basic Life Support Training Program on Quality in Cardiopulmonary Resuscitation Performance During Training and Willingness to Perform Bystander Cardiopulmonary Resuscitation: A Cluster Randomized Controlled Study. Simul Healthc. 2020 Oct;15(5):318-325. doi: 10.1097/SIH.0000000000000435. PMID 32604135
- [Background] Gurusamy KS, Aggarwal R, Palanivelu L, Davidson BR. Virtual reality training for surgical trainees in laparoscopic surgery. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD006575. doi: 10.1002/14651858.CD006575.pub2. PMID 19160288
- [Background] Aim F, Lonjon G, Hannouche D, Nizard R. Effectiveness of Virtual Reality Training in Orthopaedic Surgery. Arthroscopy. 2016 Jan;32(1):224-32. doi: 10.1016/j.arthro.2015.07.023. Epub 2015 Sep 26. PMID 26412672
- [Background] Nas J, Thannhauser J, Vart P, van Geuns RJ, Muijsers HEC, Mol JQ, Aarts GWA, Konijnenberg LSF, Gommans DHF, Ahoud-Schoenmakers SGAM, Vos JL, van Royen N, Bonnes JL, Brouwer MA. Effect of Face-to-Face vs Virtual Reality Training on Cardiopulmonary Resuscitation Quality: A Randomized Clinical Trial. JAMA Cardiol. 2020 Mar 1;5(3):328-335. doi: 10.1001/jamacardio.2019.4992. PMID 31734702
- [Background] Zheng J, Du L, Deng X, Zhang L, Wang J, Chen G. Efficacy of virtual reality techniques in cardiopulmonary resuscitation training: protocol for a meta-analysis of randomised controlled trials and trial sequential analysis. BMJ Open. 2022 Feb 11;12(2):e058827. doi: 10.1136/bmjopen-2021-058827. PMID 35149577
- [Background] Hernandez-Padilla J, Suthers F, Fernandez-Sola C, Granero-Molina J. Development and psychometric assessment of the Basic Resuscitation Skills Self-Efficacy Scale. Eur J Cardiovasc Nurs. 2016 Apr;15(3):e10-8. doi: 10.1177/1474515114562130. Epub 2014 Nov 24. PMID 25422522